CLINICAL TRIAL: NCT07208552
Title: Bishop Score Versus Cervical Length by Transvaginal Ultrasound for Predicting Success of Labor Induction Among Primigravida
Brief Title: Bishop Score vs. Cervical Length in Labor Induction
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hend ebaid mohammed kaoud, resident at the Obstetrics and Gynecology department, Assiut University
Other Study IDs: Bishop Score vs. Cervical
Record Dates: First submitted 2025-09-28; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Bishop Score; Primigravida Women; Cervical Length
Keywords: Bishop Score; primigravida women

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transvaginal Ultrasound Group (TVUS):: Participants undergo sonographic measurement of cervical length. A CL <28 mm is considered favorable for successful induction. This method provides an objective and reproducible cervical assessment.
- Bishop Score Group (BS):: Participants undergo digital vaginal examination to assign Bishop Scores. A score ≥6 is considered favorable for induction. This is the traditional method of assessing cervical readiness.

SUMMARY:
The study population consists of term primigravida women undergoing induction of labor at a tertiary care referral center in Assiut, Egypt.

DETAILED DESCRIPTION:
Participants include 88 primigravida women at ≥37 weeks of gestation, each with a singleton pregnancy in cephalic presentation. All participants present with medical or obstetric indications for induction of labor, such as post-dates, oligohydramnios, mild preeclampsia, or premature rupture of membranes. Exclusion criteria include prior uterine surgery, multiple pregnancies, malpresentation, placenta previa, vasa previa, non-reassuring fetal status at admission, or maternal infections such as active genital herpes and HIV. A carefully designed sample size calculation ensures adequate power, with a final cohort of 44 women per study arm.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy

Cephalic fetal presentation

Gestational age ≥37 weeks (confirmed by reliable dating)

Indication for induction of labor (postdate pregnancy, oligohydramnios, mild preeclampsia, premature rupture of membranes)

Exclusion Criteria:

* Previous uterine surgery (e.g., cesarean section, myomectomy)

Multiple gestation

Malpresentation

Placenta previa or vasa previa

Non-reassuring fetal heart status at admission

Active genital herpes or HIV infection

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — primigravida women
Study Population: Participants include 88 primigravida women at ≥37 weeks of gestation, each with a singleton pregnancy in cephalic presentation. All participants present with medical or obstetric indications for induction of labor, such as post-dates, oligohydramnios, mild preeclampsia, or premature rupture of membranes. Exclusion criteria include prior uterine surgery, multiple pregnancies, malpresentation, placenta previa, vasa previa, non-reassuring fetal status at admission, or maternal infections such as active genital herpes and HIV. A carefully designed sample size calculation ensures adequate power, with a final cohort of 44 women per study arm.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Rate of vaginal delivery | Within 24 hours
  The proportion of women achieving vaginal delivery after induction of labor within 24 hours of initiation.